CLINICAL TRIAL: NCT03208452
Title: The Effect of Intraoperative Magnesium Sulfate Infusion on the Occurrence of Emergence Agitation After Pediatric Ophthalmic Surgery
Brief Title: The Effect of Intraoperative Magnesium Sulfate Infusion on the Occurrence of Emergence Agitation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, LEE YEA JI, clinical professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B1605/346-002
Record Dates: First submitted 2017-06-30; First posted 2017-07-05 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Agitation,Psychomotor
MeSH Terms: conditions — Psychomotor Agitation | interventions — Magnesium Sulfate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Normal saline(NS) group (Placebo Comparator): loading 50mL of normal saline during 10minutes before starting of surgery, after starting of surgery, continuous infusion of normal saline as placebo by 0.15mg/kg/h until the end of surgery
  Interventions: Drug: Normal saline
- Magnesium group (Active Comparator): loading dose of 50mg/kg magnesium sulfate during 10minutes before starting of surgery, during the surgery, continuous infusion of magnesium sulfate by 15mg/kg/h
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — Comparing the effect of continuous infusion magnesium sulfate and normal saline in the occurrence of emergence agitation
  Other Names: 10% magnesium sulfate
  Arms: Magnesium group
Drug: Normal saline — Comparing the effect of continuous infusion magnesium sulfate and normal saline in the occurrence of emergence agitation
  Other Names: 0.9% isotonic normal saline
  Arms: Normal saline(NS) group

SUMMARY:
This study designed to evaluate the correlation between the effect of intraoperative magnesium sulfate infusion and the incidence of emergence agitation after pediatric ophthalmic surgery

DETAILED DESCRIPTION:
Emergence agitation (EA) is a frequent postoperative complication in pediatric patients after general anesthesia. There are several suggested causes of EA and pain has been considered one of them. Magnesium is an N-methyl-D-aspartate (NMDA) receptor antagonist and increasingly used as an analgesic-adjuvant. We evaluate the Pediatric Anesthesia Emergence Delirium (PAED) Scale to investigate whether the intraoperative infusion of magnesium sulfate reduces the incidence of EA in pediatric patients who undergo ophthalmic outpatient surgery.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients who are planned to operate ophthalmic surgery under general anesthesia aged 4-7 years

Exclusion Criteria:

* ASA class ≥ III
* imbalance of electrolyte
* myocardial damage or conduction abnormality on ECG
* myasthenia gravis or any other neuromuscular disease
* impaired renal function
* denial to participate in study or not be able to give informed consent

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2017-03-19 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
the incidence of emergence agitation (EA) | 15 minute interval at the post-anesthetic care unit (PACU)
  Using PAED (pediatric anesthesia emergence delirium) score, consider the score 10 or more as occuring of EA. Comparing the score between the placebo group and the intervention group for the difference of the incidence of EA.

SECONDARY OUTCOMES:
the severity of EA | 15 minute interval at the post-anesthetic care unit (PACU)
  Comparing the maximal PAED score between the placebo group and the intervention group for evaluating difference of severity of EA.

CONTACTS AND LOCATIONS:
Overall Officials: YEA JI LEE, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: No